CLINICAL TRIAL: NCT00498056
Title: A Phase IIB Test-of-Concept, Randomized, Double-Blind, Placebo-Controlled, International Clinical Trial to Evaluate the Efficacy, Safety, and Immunogenicity of a Multiclade HIV-1 DNA Plasmid Vaccine, VRC-HIVDNA016-00-VP, Followed by a Multiclade Recombinant Adenoviral Vector Vaccine, VRC-HIVADV014-00-VP, in HIV Uninfected Persons
Brief Title: Safety and Effectiveness of an HIV DNA Vaccine Followed by an HIV Adenoviral Vector Vaccine for Prevention of HIV Infection in the Americas and Africa
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); HIV Vaccine Trials Network (Network); International AIDS Vaccine Initiative (Network); US Military HIV Research Program (Network); Vaccine Research Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PAVE 100; 10500 (Registry Identifier: DAIDS ES Reigstry Number)
Record Dates: First submitted 2007-07-05; First posted 2007-07-09 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive a total of three injections of the DNA vaccine VRC-HIVDNA016-00-VP followed by one injection of the adenovirus vaccine VRC-HIVADV014-00-VP. Injections will occur at study entry and Weeks 4, 8, and 24.
  Interventions: Biological: VRC-HIVDNA016-00-VP; Biological: VRC-HIVADV014-00-VP
- 2 (Placebo Comparator): Participants will receive a total of three injections of the DNA vaccine VRC-HIVDNA016-00-VP placebo followed by one injection of the adenovirus vaccine VRC-HIVADV014-00-VP placebo. Injections will occur at study entry and Weeks 4, 8, and 24.
  Interventions: Biological: VRC-HIVDNA016-00-VP placebo; Biological: VRC-HIVADV014-00-VP placebo

INTERVENTIONS:
Biological: VRC-HIVDNA016-00-VP — DNA vaccine administered intramuscularly
  Arms: 1
Biological: VRC-HIVADV014-00-VP — Adenovirus vaccine administered intramuscularly
  Arms: 1
Biological: VRC-HIVDNA016-00-VP placebo — DNA vaccine placebo administered intramuscularly
  Arms: 2
Biological: VRC-HIVADV014-00-VP placebo — Adenovirus vaccine placebo administered intramuscularly
  Arms: 2

SUMMARY:
The development of a safe and effective vaccine is the best strategy for preventing the spread of HIV-1. The purpose of this study is to determine the safety and effectiveness of and immune responses to an HIV vaccine regimen in healthy adults at risk for HIV infection.

DETAILED DESCRIPTION:
The number of people infected by HIV-1 worldwide continues to increase. However, antiretroviral therapy is largely unavailable in low- and middle- income countries where risk of infection is very high. The development of a safe and effective vaccine to prevent HIV infection is urgently needed. This study will evaluate the effectiveness, safety, and immunogenicity of an experimental multiclade HIV vaccine, VRC-HIVDNA016-00-VP, followed by an adenovirus-vectored vaccine boost, VRC-HIVADV014-00-VP, in HIV uninfected adults. Both vaccines code for proteins from HIV subtypes A, B, and C, which together represent 75% to 85% of new HIV infections in the world. Adenoviral type 5-based vaccines have improved induction of HIV-specific CD8 cytotoxic T-lymphocyte cell responses, which correlate with lower HIV burden (viral load) and slower disease progression in primates and in HIV-1 infected people whose disease does not progress over the long term. The purpose of this study is to determine the safety and effectiveness of and immune response to a series of multiclade DNA vaccine injections followed by a booster injection of a multiclade adenovirus vaccine against HIV-1 infection in healthy adults at risk for HIV infection in North and South America, the Caribbean, and Africa.

This study will last from about 3 years to 5 years, because the length of the study depends on how quickly people enroll and how quickly during the study new HIV-1 infections occur. Study participants will be randomly assigned to receive a total of three injections of the DNA vaccine VRC-HIVDNA016-00-VP followed by one injection of the adenovirus vaccine VRC-HIVADV014-00-VP, for a total of four injections of vaccine or four injections of placebo. Injections will occur at study entry and Weeks 4, 8, and 24. Prior to the study injections, participants will have their vital signs and weight measured, and blood collection will occur. Participants will be observed in the clinic for at least 30 minutes after each injection for immediate reactions to the vaccines. At all injection visits, HIV risk-reduction counseling, HIV risk assessment, pregnancy prevention counseling, and training on how to use memory cards will also occur. For 3 to 7 days after each injection, participants will be asked to record information about injection site pain, redness, size, swelling, temperature, general well-being, and headaches on their memory cards. Additional study visits will occur on Weeks 1, 12, 28, 48, 72, 96, 120, and 144. At these visits, physical examinations, blood collection, and social impact questionnaires may also be done. Any study participants who become infected with HIV while on the study will be monitored for at least 72 weeks after diagnosis or at least 12 weeks after the study reaches its primary evaluation time point (whichever is longer). The study investigators are committed to providing access to local standard of care and treatment to those study participants who are found to be HIV-1 infected.

ELIGIBILITY:
Inclusion Criteria:

* At risk for HIV-1 sexual exposure within 24 weeks prior to study entry. More information about this criterion is available in the protocol.
* HIV uninfected within 6 weeks prior to study entry
* Willing to undergo HIV testing and counseling
* Willing to receive HIV test results
* Willing to use highly reliable method for contraception for at least the first 6 months of study

Exclusion Criteria:

* Participation in a clinical trial of another investigational product within 12 weeks prior to study entry
* Contraindication to intramuscular injections, history of bleeding disorder, or use of anticoagulant therapy in the 4 weeks prior to study entry
* Previously received an investigational HIV vaccine
* History of severe local or systemic reactogenicity to vaccines or severe allergic reactions or recurrent rash for unknown reasons in the 5 years prior to study entry
* Received an inactivated vaccine within the 2 weeks prior to study entry or of live attenuated within 4 weeks of study entry
* Received any blood products or any immunomodulatory agents within 12 weeks of study entry
* History of cancer. Participants with a history of localized squamous cell or basal cell carcinoma of the skin are not excluded.
* History of clinically significant autoimmune disease or immune deficiency syndrome
* Use of immunosuppressive medications within 24 weeks of study entry. Participants who have completed a short course of steroids more than 2 weeks prior to study entry, or using inhaled or topical steroids are not excluded.
* Seizure disorder. Participants who have had seizures with fever under the age of 2, seizures secondary to alcohol withdrawal more than 3 years prior to study entry, or a singular seizure more than 3 years ago that has not recurred or required treatment within the last 3 years are not excluded.
* Any medical condition or acute medical illness that, in the opinion of the investigator, would interfere with the study
* Pregnancy, plan to become pregnant, or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Acquisition of HIV infection, reduction in viral load in those who become infected, and adverse events (AEs) | At 26 weeks or later from study entry and from first study injection for AEs
Seroconversion with HIV RNA or HIV DNA detection, average of two viral load measurements, and AEs graded on the DAIDS AE Grading Table | Early after diagnosis of HIV infection and throughout the study for AEs

CONTACTS AND LOCATIONS:
Overall Officials: Scott M. Hammer, MD, Study Chair — Columbia University

REFERENCES:
- [Background] Esparza J, Osmanov S. HIV vaccines: a global perspective. Curr Mol Med. 2003 May;3(3):183-93. doi: 10.2174/1566524033479825. PMID 12699356
- [Background] Gaschen B, Taylor J, Yusim K, Foley B, Gao F, Lang D, Novitsky V, Haynes B, Hahn BH, Bhattacharya T, Korber B. Diversity considerations in HIV-1 vaccine selection. Science. 2002 Jun 28;296(5577):2354-60. doi: 10.1126/science.1070441. PMID 12089434
- [Background] Johnston MI, Fauci AS. An HIV vaccine--evolving concepts. N Engl J Med. 2007 May 17;356(20):2073-81. doi: 10.1056/NEJMra066267. No abstract available. PMID 17507706
- [Background] Stratov I, DeRose R, Purcell DF, Kent SJ. Vaccines and vaccine strategies against HIV. Curr Drug Targets. 2004 Jan;5(1):71-88. doi: 10.2174/1389450043490686. PMID 14738219